CLINICAL TRIAL: NCT05667441
Title: Adherence to Lifestyle Changes for Age-related Macular Degeneration
Acronym: AMD-Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: CORR foundation (Unknown)
Responsible Party: Principal Investigator, Caroline C.W. Klaver, MD, Prof. dr. C.C.W. Klaver, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL65052.078.18; MEC-2018-063 (Other: METC Erasmus MC)
Record Dates: First submitted 2022-11-21; First posted 2022-12-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration; Lifestyle; Lifestyle change; Genetic testing; Personalized risk-profiling; Gut microbiome; Coaching
MeSH Terms: conditions — Macular Degeneration | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Open label, randomized, clinical trial with 3 arms. Total study duration 2 years: intervention period for 1 year and a follow-up period of 1 year with no intervention for all study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard recommendations (Active Comparator): The first group (n=50) will receive standard care recommendations (according to Netherlands Scientific Society of Ophthalmology 2014, 'Richtlijn Leeftijdsgebonden Maculadegeneratie;): refrain from smoking; perform physical exercise regularly; increase the intake of dietary food groups such as green leafy vegetables, fruits, and fatty fish; and recommendations for supplementation with antioxidants according an established formula.
  Interventions: Combination Product: Standard lifestyle recommendations + dietary supplementation
- Standard recommendations + Risk profiling (Active Comparator): The second group (n=50) receives standard care plus personalized risk profiling. A risk scoring based on currently available literature for lifestyle and genetic risk will be used to determine personalized risks of conversion to late AMD. Individuals will be informed about their own risk profile and a personalized strategy will be communicated.
  Interventions: Combination Product: Standard lifestyle recommendations + dietary supplementation; Combination Product: Risk profiling
- Standard recommendations + Risk profiling + Additional coaching (Active Comparator): The third group (n=50) receives standard care (see 1); personalized risk profiling (see 2); and coaching. A coach will employ behavioral change techniques (BCT) to enhance adherence using motivational interviews, feedback on behavior; and focus on the advantages of following recommendations.
  Interventions: Combination Product: Standard lifestyle recommendations + dietary supplementation; Combination Product: Risk profiling; Behavioral: Coaching

INTERVENTIONS:
Combination Product: Standard lifestyle recommendations + dietary supplementation — refrain from smoking; perform physical exercise regularly; increase the intake of dietary food groups such as green leafy vegetables, fruits, and fatty fish and recommendations for supplementation with antioxidants according an established formula
Combination Product: Risk profiling — Personalized risk profiling for lifestyle and genetics.
  Arms: Standard recommendations + Risk profiling; Standard recommendations + Risk profiling + Additional coaching
Behavioral: Coaching — Coaching
  Arms: Standard recommendations + Risk profiling + Additional coaching

SUMMARY:
The AMD-Life study investigates which strategies (personalized risk-profiling including genetic testing and/or coaching) motivate AMD patients to change their lifestyle.

DETAILED DESCRIPTION:
Age-related macular degeneration is a frequent eye disease in the elderly affecting the center of retina, i.e., the macula. Despite current treatments for the wet form of this disease, it is still the most frequent cause of blindness in the Western world. The disease is the result of the interplay between genetic and environmental factors such as smoking, unhealthy diet, and lack of physical activity. The current clinical recommendations are aimed towards these lifestyle factors: a healthy diet, no smoking, regular physical exercise, and use of antioxidant supplementation. Although assumed to be low by clinicians as they feel patients find it difficult to actually alter their lifestyle, the adherence and feasibility to these recommendations in clinical ophthalmology practice is unclear. Individualizing the patients' risk of blindness and lifestyle changes, as well as coaching may positively influence adherence strategies. This pilot study aims to gain knowledge and experience in a relatively small study comparing adherence to these strategies through a healthier lifestyle. Additionally, the trial investigates blood and gut microbiome biomarkers: which molecules in blood directly relate to the supplemented nutrients as well as those related to the pathogenesis of AMD, and which biomarkers in blood and eye best correlate with supplement intake and lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Early/Intermediate AMD or unilateral late AMD with minimal vision 0.8

Exclusion Criteria:

* Participation in other intervention studies for AMD
* Living in retirement homes (difficulty in implementation of diet)
* Diagnosis of dementia (because of unreliable dietary recall)
* Persons with macular pathology other than AMD hindering appropriate grading of the macula
* Persons who are illiterate and have no independent trusted person with them to explain the informed consent form.
* Persons diagnosed with liver and kidney insufficiency.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Change in lifestyle score | 0 and 12 months: intervention phase
  Change in lifestyle as measured by online questionnaires, scale from 0-13 in which 13 represents a healthy lifestyle
Change in lifestyle score | 12 and 24 months: follow-up phase
  Change in lifestyle as measured by online questionnaires, scale from 0-13 in which 13 represents a healthy lifestyle

CONTACTS AND LOCATIONS:
Overall Officials: C.C.W. Klaver, Prof. Dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AMD-Life website with information for potential participants — http://www.maculadegeneratie.nl